CLINICAL TRIAL: NCT02906423
Title: Results From a Health System-wide Implementation of a Quality of Life Questionnaire
Status: Completed | Type: Observational
Sponsor: Allina Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 2015011
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Medical Oncology; Cardiology; Integrative Medicine; Physical and Rehabilitation Medicine; Orthopedics; Spine; Palliative Care; Pulmonary Medicine; Primary Care
Keywords: Quality of Life; Patient-Centered Care; Patient Outcome Assessment

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Allina health patients
  Interventions: Other: PROMIS-10 questionnaire

INTERVENTIONS:
Other: PROMIS-10 questionnaire — Patient completed a PROMIS-10 questionnaire

SUMMARY:
The purpose of this retrospective chart review pilot study is to research the results and scores of the QOL questionnaire implemented across Allina Health clinics. This study will investigate average QOL scores by clinical population and demographic group, the change in scores over time, and the effect of clinical interventions on QOL scores. The results will provide insight into QOL trends within different patient populations and provide guidance regarding optimal treatment plans so that Allina caregivers can positively impact patients' QOL.

DETAILED DESCRIPTION:
Quality measures, including quality of life (QOL), have become an increasingly important area of interest for health systems across the country. Systematic approaches to collect patient QOL data are needed to properly understand and act on this information. At Allina Health, the process of systematically collecting this information began in July, 2012. The information is not only collected by providers, but used to enhance the patient experience and provide patients with an active voice in their care. By considering QOL as another vital sign, Allina caregivers have an instantaneous understanding of the patient's health status and can utilize the data in real time. Additionally, by collecting this information at each visit, providers also have a longitudinal perspective of the patient's QOL and the health of the population of individuals under their care. Consequently, they can provide patients with resources and support that can have a positive impact on their health and well-being.

The purpose of this retrospective chart review pilot study is to research the results and scores of the QOL questionnaire implemented across Allina Health clinics. This study will investigate average QOL scores by clinical population and demographic group, the change in scores over time, and the effect of clinical interventions on QOL scores. The results will provide insight into QOL trends within different patient populations and provide guidance regarding optimal treatment plans so that Allina caregivers can positively impact patients' QOL.

ELIGIBILITY:
Inclusion Criteria:

* patients seen at an Allina Health outpatient facility who complete a PROMIS-10 questionnaire between July 1, 2012 and December 31, 2016.

Exclusion Criteria:

* patients who did not allow their records to be used for research purposes are not included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a retrospective chart review of up to 75,000 patients seen at an Allina Health facility who completed a Patient Reported Outcomes Measurement Information System Global Short Form (PROMIS-10) questionnaire between July 1, 2012 and December 31, 2016. Service line programs in which this questionnaire was deployed included the following: cardiac rehabilitation, heart failure, care management, physical and mental rehabilitation, integrative medicine, oncology, orthopedic, palliative care, pulmonary rehabilitation, primary care, and spine. Patients over 17 years of age who completed a PROMIS-10 questionnaire in an Allina Health clinic between July 1, 2012 and December 31, 2016 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 43000 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To investigate average baseline QOL scores by clinical population, demographic group, and across all of Allina Health. | July, 2012- December, 2014

SECONDARY OUTCOMES:
To analyze the change in QOL scores over time by clinical population and demographic group and across Allina Health. | July, 2012- December, 2014
To study the effect of programmatic clinical interventions on QOL scores by population. | July, 2012- December, 2014

CONTACTS AND LOCATIONS:
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Wolever RQ, Abrams DI, Kligler B, Dusek JA, Roberts R, Frye J, Edman JS, Amoils S, Pradhan E, Spar M, Gaudet T, Guarneri E, Homel P, Amoils S, Lee RA, Berman B, Monti DA, Dolor R. Patients seek integrative medicine for preventive approach to optimize health. Explore (NY). 2012 Nov-Dec;8(6):348-52. doi: 10.1016/j.explore.2012.08.005. PMID 23141791
- [Background] Howie L, Hirsch B, Locklear T, Abernethy AP. Assessing the value of patient-generated data to comparative effectiveness research. Health Aff (Millwood). 2014 Jul;33(7):1220-8. doi: 10.1377/hlthaff.2014.0225. PMID 25006149
- [Background] Glasgow RE, Kaplan RM, Ockene JK, Fisher EB, Emmons KM. Patient-reported measures of psychosocial issues and health behavior should be added to electronic health records. Health Aff (Millwood). 2012 Mar;31(3):497-504. doi: 10.1377/hlthaff.2010.1295. PMID 22392660